CLINICAL TRIAL: NCT05025059
Title: The EXCitE Study: Exercise During Chemotherapy in Older Women With Early-Stage Breast Cancer
Brief Title: Exercise During Chemotherapy in Older Women With Stage I-III Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0638; NCI-2021-08757 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0638 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-17; First posted 2021-08-27 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (coaching, exercise, questionnaire) (Experimental): Patients participate in one-on-one coaching sessions with a health coach QW to discuss the content offered in the program, and challenges they are currently facing in achieving their exercise goals. Patients receive a copy of the WWE workbook, wear a fitness tracker and are encouraged to achieve 150 minutes of walking per week during chemotherapy and up to 1 month after chemotherapy. Patients also participate in the Growing Stronger Strength Training Program and receive instruction manuals. They perform the initial 2 exercises 2 days per week for 4 weeks, and subsequent 2 exercises 2 days per week for the remainder of the chemotherapy course. Patients maintain exercise logs and complete questionnaires over 30-45 minutes at baseline, end of chemotherapy and at 1 month after chemotherapy.
  Interventions: Procedure: Discussion; Other: Exercise Intervention; Other: Informational Intervention; Other: Medical Device Usage and Evaluation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Discussion — Participate in coaching sessions
  Other Names: Discuss
Other: Exercise Intervention — Perform walking exercise
Other: Exercise Intervention — Perform strength exercises
Other: Informational Intervention — Receive WWE workbook and Growing Stronger Strength Training Program instruction manual
Other: Informational Intervention — Maintain exercise log
Other: Medical Device Usage and Evaluation — Wear fitness tracker
Other: Quality-of-Life Assessment — Complete questionnaires
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial evaluates the feasibility of exercise during chemotherapy in older women with stage I-III breast cancer. Previous studies have reported that exercise may reduce the chemotherapy-toxicity risk. This trial may help researchers learn if engaging in a physical activity program is feasible in patients receiving chemotherapy for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of implementing a home-based exercise intervention in older adults receiving chemotherapy for early-stage breast cancer.

SECONDARY OBJECTIVES:

I. Describe and determine the incidence of Common Terminology Criteria for Adverse Events (CTCAE) grade 3-5 toxicities overall and in three risk subgroups ("low-risk," "mid-risk" and "high-risk") determined by the Cancer and Aging Research Group-Breast Cancer (CARG-BC) tool.

II. Evaluate the accuracy of the CARG-BC tool in predicting the incidence of CTCAE grade 3-5 toxicities.

III. Determine the incidence of dose-reductions, dose-delays, treatment discontinuation and reduced-dose intensity (RDI; defined as < 85% of total dose) overall and in the three risk subgroups.

IV. Determine the incidence of hospitalizations overall and in the three risk subgroups.

V. To examine the effect of the intervention on quality of life overall and in the three risk subgroups, as assessed by the Functional Assessment of Cancer Therapy-Breast (FACT-B) and Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F).

VI. To examine the effect of the intervention on function overall and in the three risk subgroups.

VII. To examine the effects of the intervention on patient expectation and self-efficacy, as assessed by Outcomes Expectations for Exercise (OEE) and Perceived Self-Efficacy for Fatigue Self-Management (PSEFSM) respectively.

OUTLINE:

Patients participate in one-on-one coaching sessions with a health coach once a week (QW) to discuss the content offered in the program, and challenges they are currently facing in achieving their exercise goals. Patients receive a copy of the Walk with Ease Program (WWE) workbook, wear a fitness tracker and are encouraged to achieve 150 minutes of walking per week during chemotherapy and up to 1 month after chemotherapy. Patients also participate in the Growing Stronger Strength Training Program and receive instruction manuals. They perform the initial 2 exercises 2 days per week for 4 weeks, and subsequent 2 exercises 2 days per week for the remainder of the chemotherapy course. Patients maintain exercise logs and complete questionnaires over 30-45 minutes at baseline, end of chemotherapy and at 1 month after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older, female
* Histologically confirmed Stage I, II or III breast cancer (if the patient has had more than one breast cancer, then the most recent diagnosis)
* Scheduled to begin adjuvant or neoadjuvant chemotherapy regimen either as standard-of-care or on study
* English or Spanish speaking
* Able to provide written, informed consent
* Patient-assessed ability to walk and engage in moderate physical activity
* Willing and able to meet all study requirements

Exclusion Criteria:

* The presence of significant medical conditions that in the physician's judgement preclude participation in the exercise intervention

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | Up to 1 month after chemotherapy
  Will be calculated as the ratios of (a) the average number of exercise sessions completed weekly to total number of weekly targeted sessions during the period of chemotherapy (goal = 5 for walking sessions and 2 for upper-extremity exercises wearable. The mean adherence will be calculated for each patient.
Compliance | Up to 1 month after chemotherapy
  Compliance will be calculated as the ratio of the average total number of valid days (>= 10 hours /day of use) to the total number of weekly targeted days (goal = 5). The mean compliance will be calculated for each patient.
Retention | Up to 1 month after chemotherapy
  Will be assessed as the proportion of patients who enrolled in the study who complete all questionnaires and assessments at all time points.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 1 month after chemotherapy
  Chemotherapy toxicity will be measured per Common Terminology Criteria for Adverse Events version 5.0. All AEs (grade 1-5) will be captured at each follow-up visit during chemotherapy.
Geriatric assessment | Baseline up to 1 month after chemotherapy
  The Wilcoxon signed rank test will be used to assess the changes of geriatric assessment measures.
Short Physical Performance Battery (SPPB) | Baseline up to 1 month after chemotherapy
  The Wilcoxon signed rank test will be used to assess the changes physical performance (SBBP).
Quality of life questionnaires | Baseline up to 1 month after chemotherapy
  Assessed using Functional Assessment of Cancer Therapy-Breast and Functional Assessment of Chronic Illness Therapy-Fatigue. The Wilcoxon signed rank test will be used to assess the changes of quality of life measures.
Outcome Expectations for Exercise (OEE) Scale Questionnaires | Baseline up to 1 month after chemotherapy
  The Wilcoxon signed rank test will be used to assess the changes of expectations for exercise (OEE) within patient from baseline to each follow-up time point. Scale 1 (Strongly Disagree) to 5 (Strongly Agree)
Perceived Self-Efficacy for Fatigue Self-Management (PSEFSM) questionnaires | Baseline up to 1 month after chemotherapy
  The Wilcoxon signed rank test will be used to assess the changes self-efficacy for fatigue (PSEFSM) within patient from baseline to each follow-up time point. PSEFSM 35-36 is a 6-item scale that uses a 10-point response option ranging from "not at all confident" to "total confident.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Karuturi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org